CLINICAL TRIAL: NCT05851209
Title: Evaluation of Immunologic and Image Morphologic Parameters to Predict Disease Progression in Patients With Moderate Aortic Valve Stenosis
Brief Title: Biomarkers and Mechanisms of Disease Progression and Outcome of Aortic Stenosis in Humans
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Research Foundation (Other); University Bonn (Unknown); University Cologne (Unknown); Collaborative Research Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRR259 C06
Record Dates: First submitted 2023-04-14; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Aortic Stenosis; Imaging; Pathogenesis; Disease Progression; Aortic Valve Calcification; Genetics
Keywords: severe aortic stenosis; disease progression; pathogenesis of degenerative aortic stenosis; early detection; Cardiovascular magnet resonance; Transthoracal echocardiography; computertomography
MeSH Terms: conditions — Aortic Valve Stenosis; Disease Progression; Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biomarkers and mechanisms in the progression of aortic valve stenosis are sometimes not sufficiently understood. The current project will take into account image morphological and immunological aspects that predict the development of hemodynamically relevant aortic valve stenosis in order to identify high-risk patients and to develop further therapeutic options.

DETAILED DESCRIPTION:
Early recognition and management of aortic stenosis (AS) are substantial to avoid life threatening events during the clinical course. Multi-factorial complex mechanisms including fibrosis, oxidative stress, inflammation, angiogenesis, osteogenic differentiation and the effect of genetic risk variants have been proposed to be involved mechanistically in the pathogenesis of degenerative AS. It is crucial to identify the potentially involved mechanisms of AS progression in order to 1) identify patients at risk for pronounced cardiac damage and adverse outcomes that might benefit from early aortic valve replacement and 2) to discover treatment options that might slow down progression and lower adverse clinical events.

The consortium´s work has revealed that various inflammatory events play a substantial role for the onset and progression of aortic valve calcification and stenosis in cell culture and small animal experiments We hypothesize that patients with and without rapid progress to severe aortic stenosis differ in terms of genetic, immunological and imaging parameters early in the disease course, and that these parameters can be combined to create strong and reliable predictors of disease progression. Hence, we plan to assess multiple morphological, functional, genetic and immunological readouts and investigate their capacity to predict disease progression in AS in a clinical observational cohort of 938 patients with moderate AS.

This project is a working package as part of TRR259, which is a collaborative project between the three universities: Bonn, Cologne and Düsseldorf.

ELIGIBILITY:
Inclusion Criteria:

* The patient has an acquired (tricuspid) moderate aortic valve stenosis, which is the reason for regular outpatient cardiological care.
* The subject has been informed verbally and in writing about the study and has given written consent to participate in this study.
* Age > 18 years

Exclusion Criteria:

* The subject has contraindications for the performance of a magnetic resonance imaging or computed tomography (e.g., severe arrhythmias , contrast agent intolerance, a pacemaker, or severe renal insufficiency or severe renal insufficiency or claustrophobia).
* Presence of only mild or already high-grade acquired tricuspid Aortic valve stenosis
* Patient with bicuspid aortic valve
* Inability to follow the instructions of study personnel
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a moderate aortic valve stenosis
Sampling Method: Non-Probability Sample
Enrollment: 938 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
progress of aortic stenosis | 5 years
  Prevalence (number of participants) measured by transthoracic echocardiography

SECONDARY OUTCOMES:
hospitalization | 5 years
  Rate of patients (%) being hospitalized due to a progress of aortic stenois
death | 5 years
occurence of myocardial infarction | 5 years
occurence of stroke | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf; Georg Nickenig, Prof., Study Chair — University Bonn; Stephan Baldus, Prof., Study Chair — University Cologne
Locations (3):
- Germany (3):
  - University-Hospital Bonn, Bonn
  - University Hospital Cologne, Cologne
  - University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf

REFERENCES:
- See also: Website of TRR259 — https://www.trr259.uni-bonn.de/en/about-us